CLINICAL TRIAL: NCT07016750
Title: A Double-Blind Crossover of KB803 and Matched Placebo, for the Treatment and Prevention of Corneal Abrasions in Dystrophic Epidermolysis Bullosa
Brief Title: A Study Assessing KB803 Compared to Matching Placebo for the Treatment and Prevention of Corneal Abrasions in Dystrophic Epidermolysis Bullosa
Acronym: IOLITE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Krystal Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KB803-EYE-01
Record Dates: First submitted 2025-05-27; First posted 2025-06-12 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Dystrophic Epidermolysis Bullosa; DEB - Dystrophic Epidermolysis Bullosa; Recessive Dystrophic Epidermolysis Bullosa; Dominant Dystrophic Epidermolysis Bullosa
Keywords: Dystrophic Epidermolysis Bullosa; DEB; Corneal Abrasions
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica; Corneal Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KB803 (Experimental): KB803
  Interventions: Biological: KB803
- Placebo (Placebo Comparator): Vehicle
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: KB803 — Ophthalmic suspension of replication-defective, non-integrating herpes simplex virus (HSV-1) expressing the human collagen VII protein
  Arms: KB803
Drug: Placebo — Vehicle
  Arms: Placebo

SUMMARY:
KB803-EYE-01 is a Phase 3 double-blind, intra-patient crossover study, to evaluate the safety and efficacy of KB803 versus matched placebo in pediatric and adult subjects with recurrent corneal abrasions due to dystrophic epidermolysis bullosa (DEB).

DETAILED DESCRIPTION:
Subjects participating in the Sponsor's natural history study (protocol NHS) for at least 12 weeks and that meet all other eligibility criteria receive weekly ophthalmic administration of Investigational product (IP), KB803 or placebo, for the first 12-week intervention period. During the second intervention period subjects will receive the alternative IP for an additional 12 weeks. IP will be administered in the home setting by a healthcare provider. The Investigator (or designee) will contact subjects (or their parent/legal guardian) to assess for any adverse events or changes in medications, treatments, or procedures. Subjects (or their parent/legal guardian) will complete weekly symptom diaries and monthly questionnaires to document corneal abrasion symptoms and frequency and gauge overall subject (or parent/legal guardian) impressions of disease severity and disease/symptom changes during the study.

ELIGIBILITY:
Inclusion Criteria:

1. The subject and/or their parent/legal guardian must provide informed consent/assent and must be able to and willing to follow study procedures and instructions.
2. Age 6 months or older at time of informed consent/assent.
3. Confirmed diagnosis of DEB with a mutation in the COL7A1 gene.
4. Meets minimum corneal abrasion symptom frequency in the NHS study.

Exclusion Criteria:

1. Initiation of any new treatment regimen or change in treatment for ocular disease during the run-in period except for preservative free topical antibiotics or artificial tears/lubricants associated with standard of care treatment of corneal abrasions.
2. Treatment with an investigational agent or off-label ophthalmic use of an approved product during the run-in period or planned use during the study (Exceptions may be approved by the medical monitor on a case-by-case basis).
3. Any condition that, in the opinion of the Investigator, would impact the completion of all study-related assessments, interfere with the administration of study drug, and/or poses an additional risk to the subject.
4. Women who are pregnant or nursing.
5. Subject who is unwilling to comply with contraception requirements per protocol.
6. Subject is known to be noncompliant or is unlikely to comply with the requirements of the study protocol in the opinion of the Investigator.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of KB803. | 24 weeks
  Number of subjects with treatment related adverse events as assessed by CTCAE v5.
To evaluate the effect of ophthalmic KB803 versus placebo on frequency of corneal. abrasion symptoms. | 24 weeks
  Change from baseline in average number of days per month with corneal abrasion symptoms.

SECONDARY OUTCOMES:
To evaluate the effect of ophthalmic KB803 versus placebo on eye pain. | 24 weeks
  Change from baseline in average weekly eye pain score.
  Pain will be measured using a numerical scale with 0 being no hurt through 10 being the worst hurt.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Mission Dermatology Center, Rancho Santa Margarita, California
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Texas Dermatology and Laser Specialists, San Antonio, Texas